CLINICAL TRIAL: NCT02298634
Title: Biomarker for Farber Disease - An International, Multicenter, Epidemiological Protocol
Brief Title: Biomarker for Farber Disease (BioFarber)
Acronym: BioFarber
Status: Withdrawn | Type: Observational
Why Stopped: Transition into BioMetabol
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BFD 06-2018
Record Dates: First submitted 2014-10-23; First posted 2014-11-24 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Farber's Lipogranulomatosis; Ceramidase Deficiency; Hepatomegaly; Splenomegaly
Keywords: Lysosomal Storage Diseases; Lipogranulomatosis; Farber disease; Biomarker
MeSH Terms: conditions — Farber Lipogranulomatosis; Hepatomegaly; Splenomegaly; Lysosomal Storage Diseases; Erdheim-Chester Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For the development of the new biomarkers using the technique of Mass-spectometry, a blood sample will be taken via using a dry blood spot filter card. To proof the correct Farber diagnosis in those patients where up to the enrolment in the study no genetic testing has been done, sequencing of Farber will be done.
  The analyses will be done at:
  Centogene AG Am Strande 7 18055 Rostock Germany
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Patients with Farber disease or high-grade suspicion for Farber disease

SUMMARY:
Development of a new mass spectrometry-based biomarker for the early and sensitive diagnosis of Farber disease from the blood

DETAILED DESCRIPTION:
Farber disease (FD), also known as Farber's lipogranulomatosis, is an autosomal recessive lysosomal storage disease marked by a deficiency in enzyme ceramidase which causes a progressive accumulation of fatty material lipids leading to abnormalities in the joints, liver, throat, tissues and central nervous system.

FD is an extremely rare disorder, with a prevalence of less than 1/1000000. Currently only about 80 cases are reported worldwide. Disease onset is typically in early infancy but may occur later in life.

FD is caused by a mutation in the ASAH1 gene, situated on the short arm of chromosome 8. This gene codes for acid ceramidase, a lysosomal heterodimeric enzyme that hydrolyzes ceramide into sphingosine and fatty acid. To date, less than 25 distinct mutations have been identified in Farber patients, but no large deletions have yet been reported. It is inherited with an autosomal recessive pattern.

The clinical presentation of FD is characterized by the appearance of subcutaneous skin nodules, ordinarily near the joints, most often interphalangeal, wrist, elbow and ankle joints, or over points of mechanical pressure. These manifestations are very painful and lead to progressive joint stiffness, limitation of motion by contractures and finally to immobilization and deformation of joints. Also, a characteristic sign of FD is the development of a progressive hoarseness due to laryngeal involvement.

Beside these major manifestations seven phenotypes have been described which differ in severity and additional organ involvement, like the lungs, nervous system, heart and lymph nodes. Dependent on residual lysosomal ceramidase turnover, patients have a variable degree of central nervous system disease, leading to progressive neurologic deterioration. In most cases the neuronal dysfunction rather than the general physical dystrophy seems to limit the duration of FD. As well, patients with FD may die due to pulmonary disease with interstitial pneumonia.

First symptoms usually appear between the newborn period and the first birthday. Milder forms of type 3 were described with onset at 20 months of age. Clinical manifestation in type 5 of FD, dominated by neurologic deterioration, begins at 1 to 2 1/2 years of life. Patients mainly die within the first years of life, but prolonged courses in patients without severe nervous disease may also be observed.

Type 1 is the most common or classical form of this condition and is associated with the classic signs of voice, skin, and joint problems that begin a few months after birth. Developmental delay and lung disease also commonly occur. Infants born with type 1 FD usually survive only into early childhood.

Types 2 and 3 generally have less severe signs and symptoms than the other types. Affected individuals have the three classic signs and usually do not have developmental delay. Children with these types of FD typically live into mid- to late childhood.

Types 4 and 5 are associated with severe neurological problems. Type 4 usually causes life-threatening health problems beginning in infancy due to massive lipid deposits in the liver, spleen, lungs, and immune system tissues. Children with this type typically do not survive past their first year of life. Type 5 is characterized by progressive decline in brain and spinal cord (central nervous system) function, which causes paralysis of the arms and legs (quadriplegia), seizures, loss of speech, involuntary muscle jerks (myoclonus), and developmental delay. Children with type 5 FD survive into early childhood.

Types 6 and 7 are very rare, and affected individuals have other associated disorders in addition to FD.

New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity.

Therefore it is the goal of the study to identify and validate a new biochemical marker from the blood of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment.

ELIGIBILITY:
INCLUSION CRITERIA

* Informed consent will be obtained from the parents before any study related procedures.
* Patients of both gender older than 2 months
* The patient has a diagnosis of Farber disease or a high-grade suspicion for Farber disease
* High-grade suspicion present, if one or more inclusion criteria are valid:

  1. - Positive family anamnesis for Farber disease
  2. - Hoarse cry due to laryngeal involvement
  3. - Dysostosis multiplex
  4. - Painful swollen joints,
  5. - Arthritis
  6. - Hepatomegaly
  7. - Splenomegaly
  8. - Elevated urine ceramide levels
  9. - Histiocytic infiltration of liver, spleen, and lungs
  10. - Ceramidase deficiency

EXCLUSION CRITERIA

* No Informed consent from the parents before any study related procedures.
* Patients of both gender younger than 2 months
* No diagnosis of Farber disease or no valid criteria for profound suspicion of Farber disease

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Farber disease or high-grade suspicion for Farber disease
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Sequencing of the Farber disease related gene | 4 weeks
  Next-Generation Sequencing (NGS) of the ASAH1 gene will be performed. The mutation will be confirmed by Sanger sequencing.

SECONDARY OUTCOMES:
The Farber disease specific biomarker candidates finding | 24 months
  The quantitative determination of small molecules (molecular weight 150-700 kD, given as ng/μl) within a dried blood spot sample will be validated via liquid chromatography multiple reaction-monitoring mass spectrometry (LC/MRM-MS) and compared with a merged control cohort. The statistically best validated molecule will be considered as a disease specific biomarker.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Study Chair — Centogene GmbH
Locations (3):
- Children Hospital, Faculty of Medicine, Cairo University, Cairo, Egypt
- Centogene AG, Rostock, Germany
- Navi Mumbai Institute of Research In Mental And Neurological Handicap (NIRMAN), Mumbai, India

IPD SHARING:
Plan to Share IPD: Undecided